CLINICAL TRIAL: NCT03666169
Title: The Public's Response to Receiving Genetic Information Via an Electronic Platform: A Quantitative Survey
Brief Title: Receiving Genetic Information: A Quantitative Survey
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Other Study IDs: SMEC_2017-18_140
Record Dates: First submitted 2018-09-10; First posted 2018-09-11 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Whole Cohort: UK Citizens, aged 18-65 years
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey

SUMMARY:
This study will evaluate the public's response to receiving genetic information via an electronic platform. It will comprise of an internet run quantitative survey.

DETAILED DESCRIPTION:
There is currently a high prevalence of obesity in the UK. Diets personalised to an individual's genetics could help to reduce the prevalence. However, how the public will respond to this information is unknown. The use of technology is very common and could provide an accessible platform to communicate genetic results to the public. Therefore, this study will evaluate the public's response to receiving genetic information via an electronic platform.

This study will comprise of an internet run quantitative survey. The survey will be circulated using relevant websites, internet forums, emails and social media. Participants will be required to complete the survey once which will take around 10 minutes. The participants will not be required to complete the survey in a controlled setting, it may be complete wherever the participant feels comfortable. Data analysis will take place at St Mary's University.

ELIGIBILITY:
Inclusion Criteria:

UK citizens between the ages of 18 and 65 years

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: UK citizens between the ages of 18 and 65 years
Sampling Method: Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2018-10-31 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
BMI against response. | October - November 2018
  If BMI and socioeconomic status differs between participants who show a positive response to receiving genetic information to those that show a negative response.
Socioeconomic status versus response. | October - November 2018
  If socioeconomic status and socioeconomic status differs between participants who show a positive response to receiving genetic information to those that show a negative response.

IPD SHARING:
Plan to Share IPD: No